CLINICAL TRIAL: NCT03981887
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of Intravenous Nafithromycin in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Doses of Intravenous Nafithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Clinartis, LLC (Unknown); Keystone Bioanalytical, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: W-4873-105
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — nafithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nafithromycin 200 mg as IV infusion (Experimental): Nafithromycin 200 mg administered as IV infusions twice daily (q12h) over a period of 3 hours for 3 days.
  Interventions: Drug: Nafithromycin
- placebo administered as IV infusion (Placebo Comparator): Placebo administered as IV infusions twice daily (q12h) over a period of 3 hours for 3 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nafithromycin — Nafithromycin 200 mg as IV infusion
  Arms: Nafithromycin 200 mg as IV infusion
Other: Placebo — placebo administered as IV infusion
  Arms: placebo administered as IV infusion

SUMMARY:
This will be a Phase 1, randomized, double-blind, single-center, placebo-controlled study in healthy male and female adult subjects. Subjects will be randomly assigned to receive either nafithromycin or placebo by intravenous (IV) infusion based on a double-blind randomization schedule. The following treatments will be administered:

* Nafithromycin 200 mg or placebo administered as IV infusions twice daily (q12h) over a period of 3 hours for 3 days.
* Eight subjects (n=8) will receive nafithromycin and 2 subjects (n=2) will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 to ≤32 kg/m2, both inclusive.
* Stable health based on a medical history without any major pathology/surgery in the 6 months before Screening and no clinically significant physical examination findings or clinical laboratory test results
* Resting supine blood pressure of 90 to 139 mmHg (systolic) and 60 to 89 mmHg (diastolic) and a resting heart rate of 50 to 100 beats per minute at Screening and Check-in (Day -1).
* Calculated creatinine clearance ≥80 mL/min (Cockroft-Gault method) at Screening.
* Computerized 12-lead electrocardiogram (ECG) recording without signs of clinically significant pathology and showing no clinically significant deviation as judged by the investigator

Exclusion Criteria:

* Participation in another investigational drug or device study or treated with an investigational product within 30 days or 5 half-lives, whichever is longer, before study drug administration in this study.
* History/evidence of clinically relevant pathology
* History of clinically significant food or drug allergy
* Positive alcohol or urine drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
To assess safety | Day 19
  By measuring treatment emergent AEs
To assess multiple dose drug tolerability | Day 19
  By measuring treatment emergent AEs

SECONDARY OUTCOMES:
To assess plasma PK parameters profile | Day 3
  Area under the plasma concentration-time curve (AUC)
To assess plasma PK parameters profile | Day 3
  Maximum observed plasma concentration (Cmax)
To assess plasma PK parameters profile | Day 3
  Time to Cmax (Tmax)
To assess plasma PK parameters profile | Day 3
  Terminal half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States